CLINICAL TRIAL: NCT04234360
Title: Eosinophil-driven Corticotherapy for Patients Hospitalized for COPD Exacerbation: a Double-blind, Randomized, Controlled Trial
Brief Title: Eosinophil-driven Corticotherapy for Patients Hospitalized for COPD Exacerbation
Acronym: eo-Drive
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECHMPL19_0069 UF 7771; 2019-002724-33 (EudraCT Number); LIC-18-18-0374 (Other Grant/Funding Number: French DGOS PHRC National 2018)
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: This is a randomised (1:1), 2-parallel arm, double-blind trial comparing outcomes for a group of eosinophilic COPD patients (n=150) treated via corticotherapy versus a 2nd, similar group (n=150) treated via placebo. Secondarily, the same comparison (2x n=150) will be made for non-eosinophilic patients (totally excluding non-eosinophilic patients would potentially affect biomarker knowledge and subsequent care decisions, leading to bias).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, investigators / outcome assessors / care givers and study staff are blinded to eosinophil / basophil / monocyte results and treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Eosinophil count > 2%; corticotherapy (Experimental): Eosinophilic patients randomized to this arm will receive 5 days of corticotherapy.
  Interventions: Drug: 5 days of systemic corticotherapy (prednisone)
- Eosinophil count <= 2%; corticotherapy (Experimental): Non-eosinophilic patients randomized to this arm will receive 5 days of corticotherapy.
  Interventions: Drug: 5 days of systemic corticotherapy (prednisone)
- Eosinophil count > 2%; placebo (Placebo Comparator): Eosinophilic patients randomized to this arm will receive 5 days of placebo.
  Interventions: Drug: 5 days of placebo
- Eosinophil count <= 2%; placebo (Placebo Comparator): Non-eosinophilic patients randomized to this arm will receive 5 days of placebo.
  Interventions: Drug: 5 days of placebo

INTERVENTIONS:
Drug: 5 days of systemic corticotherapy (prednisone) — Patients randomized to this arm will receive 40 mg prednisone per os per day for 5 days. Other aspects of standard, recommended care (e.g. antibiotherapy) are respected.
  Arms: Eosinophil count <= 2%; corticotherapy; Eosinophil count > 2%; corticotherapy
Drug: 5 days of placebo — Patients randomized to this arm will receive an appropriate placebo per os for 5 days. Other aspects of standard, recommended care (e.g. antibiotherapy) are respected.
  Arms: Eosinophil count <= 2%; placebo; Eosinophil count > 2%; placebo

SUMMARY:
The primary objective of this study is to compare treatment failure rates between a group of eosinophilic (eosinophilia > 2% on day 1 of hospitalization) patients hospitalised for a COPD exacerbation treated via corticotherapy versus a similar group treated via placebo.

Secondarily, treatment failure rates will also be compared between a group of non-eosinophilic patients hospitalised for a COPD exacerbation treated via corticotherapy versus a similar group treated via placebo. Study arms will also be compared for additional aspects of efficacy and safety:

* speed of recovery during the initial hospitalization;
* corticosteroid side effects / induced comorbidities;
* changes in symptoms and episodes of exacerbation;
* pulmonary function, oxygen use and ventilation;
* patient trajectories and resource use (e.g. survival, consults, episodes of hospitalization, medications);
* drug consumption (especially as relates to COPD management, exacerbations and induced comorbidities);
* health status, quality of life, activity/disability;
* patient safety / adverse events in general.

Eosinophilia thresholds optimizing the prediction of corticosteroid response and COPD outcomes will be re-evaluated. The relationships between corticosteroid response and key biomarkers (e.g. infectious groups) will be thoroughly explored, including within eosinophil strata. Potential gender subgroups differences will also be evaluated.

Finally, in prevision of further exploratory studies, a biological collection and an imaging library will be created in association with this protocol. The biological collection will be used to explore the genetic basis and physiology linked with treatment response, gender and patient trajectories. The image library will be used as a platform for the exploration of new imaging markers developed, for example, via machine learning and affiliated techniques.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to a participating hospital (ward, ICU or emergency services) for an acute COPD exacerbation
* For patients with known COPD: COPD defined according to GOLD 2018 criteria: (1) Post-bronchodilator FEV1/FVC < 70% of predicted values; (2) > 10 pack years smoking history
* For incident COPD cases with no spirometric history: symptoms and exposure according to GOLD 2018 report will be considered for the diagnosis, but if the spirometric diagnosis is not confirmed during follow-up, then the patient will be excluded
* Signed consent has been obtained, or the appropriate emergency procedure (under French law) allows enrolment
* Subjects must be covered by public health insurance
* Patient available for 3 months of follow-up. Subjects must be able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* Subject unable to read or write; language barrier
* Subject who is in a dependency or employment with the sponsor or investigator
* Pregnancy or lactation
* Patients who are prisoners or under other forms of judicial protection
* Patients under any kind of guardianship
* The patient has already participated in the present protocol
* The patient is participating in another interventional study or has done so in the past 3 months
* The patient is in an exclusion period determined by a previous study
* The patient has been taking long-term systemic corticosteroids for longer than 1 month prior to inclusion
* The patient has already received > 1 mg/kg of systemic corticotherapy in the past 48h
* Intubated-ventilated patient
* Administration of oral experimental drug is impossible
* Cancer within the last 12 months
* Current diagnosis of Asthma
* T2-inflammation targeting biologics (Benralizumab, reslizumab, mepolizumab, dupilumab) treatment
* Admitted for any other reason including, but not limited to, pulmonary embolism, pneumothorax, heart failure
* Known allergy to corticosteroids
* Consideration of a potential negative drug interaction with corticosteroids (at the investigator's discretion)
* White blood cell formula already performed and distributed to implicated teams
* Directives for limitation-of-care ("LATA" in French) already established
* SARS-Cov2 positive test carry out during the COPD exacerbation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-10-12 (Estimated); Study Completion 2025-01-12 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 3 months
  Treatment failure for the primary outcome is defined according to Niewoehner et al. (1999) as death from any cause or need for intubation and mechanical ventilation, readmission due to COPD, or intensification of pharmacologic therapy (defined as the prescription of open-label systemic glucocorticoids, high-dose inhaled glucocorticoids (more than eight puffs per day of triamcinolone acetonide or its equivalent), theophylline, or any combination of these three therapies) at three months. In addition, an investigator meeting determined additional components of treatment failure that should be added to Niewoehner's definition in order to bring it up-to-date :
  * Initiation of non-invasive ventilation for >24h after first treatment administration
  * Transfer to intensive care or indication for a transfer to intensive care. Incident limitations-of-care that can affect treatment failure should also be carefully noted.

SECONDARY OUTCOMES:
The speed of initial recovery: Time elapsed before showing signs of improvement | During initial hospitalization (expected maximum of 28 days)
The speed of initial recovery: Time elapsed in acidosis/hypercapnia | During initial hospitalization (expected maximum of 28 days)
The speed of initial recovery: Time elapsed before meeting pre-defined discharge criteria | During initial hospitalization (expected maximum of 28 days)
  Time elapsed before meeting pre-defined discharge criteria (acidosis has normalized, symptoms have returned to manageable levels, the patient is capable of performing minimal daily activities).
Presence /absence of comorbidities or steroid side effects: glycemia | During initial hospitalization (expected maximum of 28 days)
Presence /absence of comorbidities or steroid side effects: glycemia | 1 month
Presence /absence of comorbidities or steroid side effects: glycemia | 3 months
The occurrence of new or worsened diabetes/hyperglycemia | Throughout the study (3 months)
Body mass index | Baseline (day 0)
Body mass index | At hospital discharge (expected maximum of 28 days)
Body mass index | 1 month
Body mass index | 3 month
Hospital anxiety and depression scale (HAD) | baseline (day 0)
  The HAD results in a score ranging from 0 (low anxiety or depression) to 21 (strong anxiety or depression).
Hospital anxiety and depression scale (HAD) | 3 months
  The HAD results in a score ranging from 0 (low anxiety or depression) to 21 (strong anxiety or depression).
The occurrence of any other potentially corticosteroid-induced comorbidities throughout the study | Throughout the study; 3 months
Episodes of pneumonia | Throughout the study; 3 months
  Beginning and end dates of episodes.
Episodes of infection | Throughout the study; 3 months
  Beginning and end dates of episodes.
Episodes of mild exacerbation. | Throughout the study; 3 months
  Episodes of exacerbation will be recorded (date of start/finish for each episode) throughout the study.
  Exacerbation severity is determined (GOLD 2018) as follows:
  * mild: treated with short acting bronchodilators (SABDs) only,
  * moderate: treated with SABDs plus antibiotics and/or oral corticosteroids,
  * severe: patient required hospitalization or visits the emergency room.
Episodes of moderate exacerbation. | Throughout the study; 3 months
  Episodes of exacerbation will be recorded (date of start/finish for each episode) throughout the study.
  Exacerbation severity is determined (GOLD 2018) as follows:
  * mild: treated with short acting bronchodilators (SABDs) only,
  * moderate: treated with SABDs plus antibiotics and/or oral corticosteroids,
  * severe: patient required hospitalization or visits the emergency room.
Episodes of severe exacerbation. | Throughout the study; 3 months
  Episodes of exacerbation will be recorded (date of start/finish for each episode) throughout the study.
  Exacerbation severity is determined (GOLD 2018) as follows:
  * mild: treated with short acting bronchodilators (SABDs) only,
  * moderate: treated with SABDs plus antibiotics and/or oral corticosteroids,
  * severe: patient required hospitalization or visits the emergency room.
Forced expiratory volume in 1 second (litres) | At hospital discharge (expected maximum of 28 days)
Forced expiratory volume in 1 second (litres) | 3 months
Forced expiratory volume in 1 second (% predicted) | At hospital discharge (expected maximum of 28 days)
Forced expiratory volume in 1 second (% predicted) | 3 months
Forced vital capacity (litres) | At hospital discharge (expected maximum of 28 days)
Forced vital capacity (litres) | 3 months
Forced vital capacity (% predicted) | At hospital discharge (expected maximum of 28 days)
Forced vital capacity (% predicted) | 3 months
Residual volume (litres) | At hospital discharge (expected maximum of 28 days)
Residual volume (litres) | 3 months
Residual volume (% predicted) | At hospital discharge (expected maximum of 28 days)
Residual volume (% predicted) | 3 months
Total lung capacity (litres) | At hospital discharge (expected maximum of 28 days)
Total lung capacity (litres) | 3 months
Total lung capacity (% predicted) | At hospital discharge (expected maximum of 28 days)
Total lung capacity (% predicted) | 3 months
Oxygen needs (litres/min) during initial hospitalisation | At hospital discharge (expected maximum of 28 days)
Mode of pre-hospitalization living arrangements | Baseline (day 0)
  At home, rehabilitation centre, assisted living centre, or other
Hospital discharge modality | At hospital discharge (expected maximum of 28 days)
  At home, rehabilitation centre, assisted living centre, or other
Episodes of hospitalization | Throughout the study; 3 months
  Episodes of hospitalization, distinguishing emergency department, intensive care, intermediate care and ward stays, will be recorded throughout the study .
Episodes of emergency department use | Throughout the study; 3 months
Episodes of intensive care | Throughout the study; 3 months
Consults | Throughout the study; 3 months
  The number of consults and rehabilitation/therapy sessions in relation to COPD/respiratory symptoms (or not) will be tracked.
The cumulative days alive and event-free | Throughout the study; 3 months
  The cumulative days alive and event-free (free from hospitalization, exacerbation, ventilation, oxygen use, pneumonia or infection)
Mortality/survival | Throughout the study; 3 months
Medications | Throughout the study; 3 months
  Drug consumption episodes (including vaccines) will be recorded throughout the study and linked to COPD exacerbations, COPD maintenance therapy or corticosteroid-induced side effects as appropriate.
VAS scale for coughing | Every morning during hospitalization (expected maximum of 28 days)
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for coughing | 1 month
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for coughing | 3 months
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for dyspnoea | Every morning during hospitalization (expected maximum of 28 days)
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for dyspnoea | 1 month
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for dyspnoea | 3 months
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for sputum production | Every morning during hospitalization (expected maximum of 28 days)
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for sputum production | 1 month
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for sputum production | 3 months
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for sleep perturbation | Every morning during hospitalization (expected maximum of 28 days)
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for sleep perturbation | 1 month
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for sleep perturbation | 3 months
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for anxiety | Every morning during hospitalization (expected maximum of 28 days)
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for anxiety | 1 month
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
VAS scale for anxiety | 3 months
  Patient reported, separate visual analogue scales (VAS) for coughing, dyspnoea (at rest), sputum production, sleep perturbation and anxiety.
  VAS scales range from 0 (absence of symptoms) to 10 (strongest possible symptoms imaginable).
The Breathlessness, Cough and Sputum Scale | Baseline (day 0)
  Symptoms are evaluated on a 5-point Likert-type scale ranging from 0 to 4, with higher scores indicating more severe symptoms.
The Breathlessness, Cough and Sputum Scale | On hospital discharge (expected maximum of 28 days)
  Symptoms are evaluated on a 5-point Likert-type scale ranging from 0 to 4, with higher scores indicating more severe symptoms.
The Breathlessness, Cough and Sputum Scale | 1 month
  Symptoms are evaluated on a 5-point Likert-type scale ranging from 0 to 4, with higher scores indicating more severe symptoms.
The Breathlessness, Cough and Sputum Scale | 3 months
  Symptoms are evaluated on a 5-point Likert-type scale ranging from 0 to 4, with higher scores indicating more severe symptoms.
The modified medical research council (mMRC) dyspnoea scale | Baseline (day 0)
  Scores range from 0 (none) to 4 (very severe).
The modified medical research council (mMRC) dyspnoea scale | 3 months
  Scores range from 0 (none) to 4 (very severe).
The COPD assessment test | Baseline (day 0)
  Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
The COPD assessment test | 1 month
  Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
The COPD assessment test | 3 months
  Scores range from 0-40 with higher scores indicative of greater COPD impact on health status.
The Euroqol (EQ-5D-5L) questionnaire | Baseline (day 0)
  The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The Euroqol (EQ-5D-5L) questionnaire | 1 month
  The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The Euroqol (EQ-5D-5L) questionnaire | 3 months
  The descriptive system has five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each described by five levels of intensity ("no problems", "slight problems", "moderate problems", "severe problems" and "extreme problems or complete inability"). This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The St George Respiratory Questionnaire | 3 months
  Scores range from 0 to 100, with higher scores indicating more limitations.
Six minute walking tests | 1 month (optional)
Six minute walking tests | 3 months
The DIRECT questionnaire | 3 months
  DIRECT: Disability related to Chronic Obstructive Pulmonary Disease (COPD) tool The DIRECT questionnaire provides a score ranging between 0 and 34, with higher values indicating higher levels of disability.

OTHER OUTCOMES:
Blood differential | Baseline (day 0)
Blood differential | day 2
Blood differential | On hospital discharge (expected maximum of 28 days)
Blood differential | 1 month
Blood differential | 3 months
C reactive protein | Baseline (day 0)
C reactive protein | On hospital discharge (expected maximum of 28 days)
Sputum bacteriological analysis (or nasal swab if no sputum) | Baseline (day 0)
Nasal swab virology | Baseline (day 0)
Computed tomography scan of lungs: presence/absence of consolidation | Baseline (day 0); optional
Computed tomography scan of lungs: presence/absence of consolidation | 3 months; optional
Computed tomography scan of lungs: % emphysema | Baseline (day 0); optional
Computed tomography scan of lungs: % emphysema | 3 months; optional

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud BOURDIN, Principal Investigator — a-bourdin@chu-montpellier.fr
Locations (21):
- France (21):
  - CHU Amiens, Amiens
  - CHU Brest - Hôpital Caval Blanche, Brest
  - Clinique du Parc, Castelnau-le-Lez
  - Centre hospitalier intercommunal de Créteil, Créteil
  - CH Libourne, Libourne
  - CHRU Lille, Lille
  - Hospice Civils de Lyon, Lyon
  - APHM - Hôpital Nord, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nancy, Nancy
  - CHU Nîmes, Nîmes
  - APHP - Hopital Européen Georges Pompidou, Paris
  - APHP - Hôpital BICHAT, Paris
  - APHP - Hôpital Cochin, Paris
  - APHP - Hôpital Universitaire Pitié-Salpétrière, Paris
  - CHU Bordeaux - Hôpital Haut Lévêque, Pessac
  - CHU Reims, Reims
  - CH Roubaix, Roubaix
  - CHRU Strasbourg, Strasbourg
  - Hôpital Larrey CHU Toulouse, Toulouse
  - Hôpital Nord Franche-Comté, Trévenans

IPD SHARING:
Plan to Share IPD: Yes
The general goal is to make the study data available to interested researchers as well as to provide proof of transparency for the study. Data (and an accompanying data dictionary) will be de-identified and potentially further cleaned or aggregated as the investigators deem necessary to protect participant anonymity.
  Data will be made available to persons who address a reasonable dataset request to the sponsor coordinating team (c/o Dr Carey Suehs, Department of Medical Information, Hôpital La Colombière, 39 avenue Charles Flahault, 34295 Montpellier Cedex 5, France).
  In accordance with French law, dataset usage requests must by approved by the French CNIL (Commission Nationale de l'Informatique et des Libertés : https://www.cnil.fr/professionnel) prior to access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Datasets (and accompanying analytic code) can be requested after the publication process has been completed.
  The protocol, SAP and information materials will be made available in real-time (in as much as possible) on the study website at the Open Science Framework.
Access Criteria: The conditions under which members of the public will be granted access to datasets are:
  * The data will be used/examined in a not-for-profit manner;
  * The data will not be used in an attempt to identify a participant or group of participants;
  * The user does not work for a private insurance company;
  * The data will not be used in support of any kind of private insurance policy or health penalties;
  * The data will be used/examined for the advancement of science/teaching while respecting participant/patient privacy and rights;
  * The user will state why they wish to access the data.
  * The appropriate CNIL approval has been obtained by the user.
URL: https://osf.io/9j7uk/

REFERENCES:
- [Background] Suehs CM, Zysman M, Chenivesse C, Burgel PR, Couturaud F, Deslee G, Berger P, Raherison C, Devouassoux G, Brousse C, Roche N, Molimard M, Chinet T, Devillier P, Chanez P, Kessler R, Didier A, Martinat Y, Le Rouzic O, Bourdin A. Prioritising outcomes for evaluating eosinophil-guided corticosteroid therapy among patients with acute COPD exacerbations requiring hospitalisation: a Delphi consensus study. BMJ Open. 2020 Jul 1;10(7):e035811. doi: 10.1136/bmjopen-2019-035811. PMID 32611741
- See also: eo-Drive on the Open Science Framework — https://osf.io/9j7uk/